CLINICAL TRIAL: NCT05490498
Title: Exploration of Breast Milk by Culture Through "Microbial Culturomics" and by Targeted Metagenomics Through 16S Ribosomal RNA Gene Sequencing. Influence on the Development of Early and Late Neonatal Sepsis in Infants Under Three Months of Age.
Brief Title: Study of the Breast Milk Microbiota and Its Influence on the Development of Early and Late Neonatal Bacterial Sepsis Under Three Months of Age.
Acronym: MINEOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-11; ID-RCB (Other: 2021-A01671-40)
Record Dates: First submitted 2022-08-03; First posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Neonatal Sepsis
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breastfeeding mother (Experimental): Breastfeeding mother with infants between 1 and 89 days of age who presented with suspected neonatal bacterial sepsis due to the presence of a fever.
  Interventions: Other: Collection of breast milk

INTERVENTIONS:
Other: Collection of breast milk — Collection of breast milk through a sterilized breastfeeding device. Once the collection is completed, the milk will be transferred to a sterile jar provided in a dedicated survey package for transport to the laboratory.

SUMMARY:
Breast milk contains many microorganisms including bacteria that are beneficial to health (probiotics), but also bacteria that are generally considered pathogenic.

Several studies have described an increased risk of infections due to pathogenic germs in breast milk in premature newborns whose digestive system is immature and whose digestive flora is modified by repeated antibiotic treatments.

However, a breastfed baby is better protected against infectious diseases than a bottle-fed baby. The objective of this study is to define the breast milk microbiota of infants with confirmed early or late neonatal bacterial infection compared to the breast milk microbiota of infants with no evidence of bacterial infection. For that purpose, an exploration will be performed using the principle of "Microbial Culturomics" and targeted metagenomics (16S ribosomal RNA gene sequencing).

ELIGIBILITY:
Inclusion Criteria:

Breastfeeding mothers of infants:

* Aged 1 to 89 days consulting in hospitals in the Marseille area (Assistance Publique des Hôpitaux de Marseille: Hôpital de la Timone-enfants and Hôpital Nord),
* Suspected neonatal bacterial infection due to the presence of fever (rectal or axillary temperature > 38°C),
* In whom bacteriological samples have been taken (cerebrospinal fluid, joint fluid, blood cultures, urine),
* Patients affiliated or benefiting from a social security system.

Exclusion Criteria:

* Exclusive formula milk feeding
* Opposition of legal guardians
* No bacteriological sample to prove infant infection
* No confirmation of fever by standardized method
* Opposition to participating in the study
* Neonatal hospitalization > 48 hours for management of prematurity.
* Severe congenital malformations in the infant.
* Antibiotic treatment for a concomitant bacterial infection in the infant.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Breastfeeding mothers
Enrollment: 75 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2024-07-12 (Estimated); Study Completion 2024-12-12 (Estimated)

PRIMARY OUTCOMES:
Description of bacterial carriage of breast milk | 18 months
  Identify the bacterial carriage of breast milk of infants with neonatal sepsis. Microbial anlaysis of mother's milk from baby with neonatal sepsis.

SECONDARY OUTCOMES:
Comparison of breast milk of infants with neonatal sepsis to infants without neonatal sepsis. | 18 months
  Compare the bacterial carriage (type of germs found) of the breast milk of infants with neonatal sepsis to breast milk of infants with fever for another cause (virus, non identified germ)
Comparison of milk germs to children's germs. | 18 months
  Compare the germs found in the breast milk of each mother-infant pair with a bacterial infection with the germs identified in the infant.
Comparison of microbiota profiles in breast milk | 18 months
  Compare the bacterial composition of the breast milk of mother-infant pairs with the same germ (germ infecting the child identical to the germ identified in the mother's milk) versus mother-infant pairs with a different germ in the milk (no germ found in the child when a germ was identified in the breast milk, or germ infecting the child different from the germ identified in the mother's milk).

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — ASSISTANCE PUBLIQUE DES HOPITAUX DE MARSEILLE
Locations (1):
- Hopital de la Timone, Marseille, France

IPD SHARING:
Plan to Share IPD: No